CLINICAL TRIAL: NCT02908828
Title: Effect of Copepod Oil Supplementation (Calanus Finmarchicus) on Endurance and VO2max in Healthy Obese Subjects
Brief Title: Calanus Oil Supplementation and Maximal Oxygen Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: University of Tromso (Other); Calanus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015/2303
Record Dates: First submitted 2016-09-14; First posted 2016-09-21 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Healthy
Keywords: Biological Products/therapeutic use; Copepoda; Dietary Supplements; Fish Oils; Fatty Acids, Omega-3; Oxygen Consumption; Calanus; Maximal oxygen uptake; Zooplankton

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calanus oil (Experimental): 4 capsules of 500 mg Calanus oil once every day
  Interventions: Dietary Supplement: Calanus oil
- Placebo (Placebo Comparator): 4 capsules of 500 mg dietary oil once every day
  Interventions: Dietary Supplement: placebo dietary oil

INTERVENTIONS:
Dietary Supplement: Calanus oil
  Arms: Calanus oil
Dietary Supplement: placebo dietary oil
  Arms: Placebo

SUMMARY:
Copepod oil is extracted from the marine copepod Calanus finmarchicus, the dominant plankton species in the marine food web in the Norwegian Sea. Copepods constitute the largest renewable and harvestable resource in the Norwegian Sea and adjacent waters, and it is now developed knowledge and technology for sustainable harvesting of this "new" resource. The purpose of this study is to investigate whether Calanus copepod oil supplementation has an equivalent effect on maximal oxygen uptake in humans to that seen in experimental studies in mice.

ELIGIBILITY:
Inclusion Criteria:

* in good health
* Body mass index (BMI) between 18,5 and 29,9

Exclusion Criteria:

* Medical condition limiting VO2max (COPD or asthma).
* diagnosed coronary artery disease
* Any other significant medical condition
* medication effecting exercise capacity (e.i. betablockers)
* Pregnancy
* Participation in other clinical trials
* Shellfish allergies
* Systolic blood pressure > 170 mmHG, or diastolic BP > 105 mmHG.
* contraindications for maximal exercise testing

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
maximal oxygen uptake (VO2max) | 6 months
  Measured with indirect calorimetry at a treadmill (running/walking) with gradually increasing work load until exhaustion. After 10-15 min with warmup at 70% of maximal heart rate, work load will be increased every 1-2 minute and the changes maximal oxygen uptake (VO2) will be recorded automatically.

SECONDARY OUTCOMES:
Body composition (InBody, Japan) | 6 months
Self-reported physical activity | 6 months
  assessed with International Physical Activity Questionnaire (IPAQ) short version

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisløff, phd prof, Study Director — Norwegian University of Science and Technology; Trine Karlsen, phd, Principal Investigator — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - Institutt for Medisinsk Biologi, UiT Norges arktiske universitet, Tromsø
  - KG Jebsen-senter for Hjertetrening, NTNU, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided